CLINICAL TRIAL: NCT04961814
Title: Gastric Ultrasound Assessment of Two Preoperative Fasting Regimens in Pediatric Patients: a Randomized Clinical Trial.
Brief Title: Preoperative Pediatric Fasting Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Raafat Elghamry, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB No: 34601/4/21
Record Dates: First submitted 2021-06-05; First posted 2021-07-14 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- standard fasting (Active Comparator): preoperative fasting according to 6-4-2 regimen then preoperative bedside gastric ultrasound assessment will be done
  Interventions: Other: standard fasting
- liberal fasting (Experimental): preoperative fasting according to 6-4-0 regimen then preoperative bedside gastric ultrasound assessment will be done
  Interventions: Other: liberal fasting

INTERVENTIONS:
Other: liberal fasting — preoperative fasting according to 6-4-0 regimen then qualitative and quantitative preoperative gastric ultrasound assessment will be done to evaluate the proportion of patients with risky stomach
  Arms: liberal fasting
Other: standard fasting — preoperative fasting according to 6-4-2 regimen then qualitative and quantitative preoperative gastric ultrasound assessment will be done to evaluate the proportion of patients with risky stomach
  Arms: standard fasting

SUMMARY:
The presence of gastric contents makes an aspiration event more likely , and as a result, preoperative fasting guidelines are designed to provide adequate time for gastric emptying in patients undergoing surgery. this study will be conducted to assess the gastric volume and content with the help of ultrasound in fasted pediatric patients scheduled for elective surgeries

DETAILED DESCRIPTION:
it is unknown how many patients have gastric volumes that place them at increased risk of aspiration despite adequate fasting.

There is a growing interest in the use of bedside ultrasonography to assess gastric content and volume. It has been suggested that the gastric antrum in particular can be assessed reliably by sonography.

hence, this study will be conducted to assess the gastric volume and content with the help of ultrasound in fasted pediatric patients scheduled for elective surgeries which will help to detect accuracy of preoperative fasting hours.

ELIGIBILITY:
Inclusion Criteria:

* paediatric patients aged 6-12 years old
* ASA physical status I and II
* scheduled for elective surgeries
* the anticipated duration of 30-60 min

Exclusion Criteria:

* parents' refusal
* overweight or obesity
* expected difficult airway management
* increased abdominal pressure
* diabetes mellitus
* congenital diseases
* GERD or esophageal disease
* uncooperative patients,
* mental retardation or neurological disease
* upper airway surgeries.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a risky stomach. | immediately preoperative
  bedside ultrasound to estimate the gastric volume in milliliter

SECONDARY OUTCOMES:
gastric content quality | immediately preoperative
  bedside ultrasound to determine the nature of gastric content (solid or fluid)
fasting hours | the new preoperative fasting (6 hours for solids, 4 hours for milk, non-clear fluid or light breakfast, and 0 hours for clear fluids)
  actual and prescribed preoperative fasting
type of last meal | last meal within 24 hours preoperative
  last meal (heavy solid,light solid,non clear fluid,or clear fluid)
episodes of gastric regurgitation, vomiting , aspiration | during induction or emergence from anesthesia (within 30 minutes)
  incidence of regurgitation, vomiting , aspiration if regurgitation happened patients will be followed up postoperative clinically and radiologically
gastric volume | immediately preoperative (within 30 minutes)
  quantitative gastric ultrasound assessment (gastric volume, volume/weight, antral cross sectional area)
parents satisfaction | after PACU discharge (within 2 hours postoperative)
  parents' satisfaction is evaluated using a 5-point Likert scale
cancellation | decision will be taken within 30 minutes preoperative
  rate of surgery cancellation
adverse events | preoperative or postoperative
  adverse events related to fasting duration

CONTACTS AND LOCATIONS:
Overall Officials: Mona R Elghamry, MD, Principal Investigator — Tanta University, Faculty of Medicine
Locations (1):
- Tanta University, Faculty of Medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
statistics of demographic data, gastric volume, fasting hours, type of last meal, episode of gastric regurgitation
Supporting Information: SAP
Time Frame: the IPD will be shared after finishing and publication of the study and it will be available for 6 months
Access Criteria: the IPD will be available for scientific research only upon e-mail request which will be sent to principal investigator (drmonagh19802000@gmail.com)

REFERENCES:
- [Derived] Elghamry MR, Elkeblawy AM, Alshawadfy AM, Ramadan KM. Gastric ultrasound assessment of two preoperative fasting regimens in pediatric patients: A randomized clinical trial. Acta Anaesthesiol Scand. 2025 Jan;69(1):e14566. doi: 10.1111/aas.14566. PMID 39711127